CLINICAL TRIAL: NCT05992571
Title: The Impact of Acute Oral Ketone Monoester Supplementation on Resting-state Brain Connectivity in Adults With Memory Complaints
Brief Title: Oral Ketone Monoester Supplementation and Resting-state Brain Connectivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Alzheimer's Society of Brant, Haldimand Norfolk, Hamilton Halton (Unknown)
Responsible Party: Principal Investigator, Jeremy Walsh, Assistant Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: rs-KME
Record Dates: First submitted 2023-06-07; First posted 2023-08-15 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Cerebrovascular Function; Cognition
Keywords: Beta-hydroxybutyrate (β-OHB); cerebral blood flow; cognition; brain connectivity

STUDY DESIGN:
Intervention Model Description: A randomized double-blind placebo-controlled crossover design will be used to test two conditions. Participants will consume 60 mL of: 1) a drink containing a ketone monoester supplement ([R]-3-hydroxybutyl [R]-3-hydroxybutyrate; 0.3 g β-OHB/kg body weight); and 2) a taste-matched calorie-free inert placebo drink.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Single dose of a taste-matched calorie-free placebo
  Interventions: Other: Placebo
- β-OHB (Experimental): Single dose of a ketone monoester ([R]-3-hydroxybutyl [R]-3-hydroxybutyrate; 0.6 g β-OHB/kg body weight)
  Interventions: Dietary Supplement: β-OHB

INTERVENTIONS:
Other: Placebo — Ingestion of a taste-matched calorie-free placebo drink followed by 90 minutes of rest.
  Arms: Placebo
Dietary Supplement: β-OHB — Ingestion of a high dose [R]-3-hydroxybutyl [R]-3-hydroxybutyrate (0.6 g β-OHB/kg body weight) followed by 90 minutes of rest.
  Arms: β-OHB

SUMMARY:
People who report subjective memory complaints have a greater risk of developing dementia. Memory issues may be an early warning sign of dysfunctional cerebral glucose metabolism and cerebral blood flow. Interventions that can restore cerebral metabolism and enhance cerebral blood flow may protect against conversion to dementia. Exogenous ketone supplements have been shown rapidly improves brain network function in young adults. Further, infusion studies demonstrate that ketone bodies enhance cerebral blood flow in cognitively normal adults. Whether acute ketone monoester supplementation can improve brain function in adults with subjective memory complaints is currently unknown.

This study will investigate the effects of a single ketone monoester dose on resting-state functional connectivity in the default mode network and resting cerebral blood flow in adults with subjective memory complaints.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 55 and 70
* presence of subjective memory complaints as determined by the Prospective- Retrospective Memory Questionnaire
* cognitively normal, e.g. score ≥26 on the Montreal Cognitive Assessment

Exclusion Criteria:

* Presence of obesity (body mass index > 30 kg/m^2)
* Presence of known cardiovascular disease
* Presence of type 2 diabetes
* History of cardiovascular events requiring hospitalization in the past 3 years (e.g., heart attack, stroke)
* History of concussion(s) with persistent symptoms
* Currently following a ketogenic diet and/or taking ketone body supplements
* Diagnosis of any form of Alzheimer's disease or dementia

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Brain network connectivity | 90 minutes
  Functional connectivity of the default mode network (DMN) is measured via functional MRI. Changes in BOLD signal in each region are determined by independent component analysis and then functional connectivity is measured as a Pearson correlation (r) between the neural regions comprising the DMN and transformed into a z score.
Cerebral blood flow | 90 minutes
  Sum of blood flow in the internal carotid and vertebral arteries via phase contrast MRI in ml/min.

SECONDARY OUTCOMES:
Working memory | 90 minutes
  Computer battery to assess working memory (n-back test) based on N2 reaction time
Executive function | 90 minutes
  Computer battery to assess executive function (Stroop test) based on Stroop Cost (reaction times to incongruent stimuli minus congruent stimuli).
Attention and working memory | 90 minutes
  Computer battery to assess working memory (digit symbol substitution task) based on the number of correct responses in 120 seconds.

OTHER OUTCOMES:
Mean arterial pressure | 90 minutes
  Automated blood pressure cuff measurement of brachial artery pressure in mmHg.
Plasma beta-hydroxybutyrate | 90 minutes
  Measured via finger capillary samples in mM

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Walsh, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual patient data (de-identified) with researchers upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Anyone who wishes to access the data.